CLINICAL TRIAL: NCT03854669
Title: Does Pain Reporting Accuracy Relates to the Intensity of Acute Post-operative Pain and Analgesic Drug Consumption?
Brief Title: Experimental Pain Reporting Accuracy and Clinical Post-operative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Principal Investigator, Tal Honigman, Principal Investigator, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMC-18-0082-CTIL
Record Dates: First submitted 2019-02-13; First posted 2019-02-26 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Surgical Procedure, Unspecified; Pain, Postoperative; Ear, Nose, and Throat (ENT) Disease
Keywords: Acute post-operative pain; Clinical pain variability; Experimental pain variability; FAST; pain reporting accuracy
MeSH Terms: conditions — Pain, Postoperative; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessing pain reporting accuracy (Experimental): Subjects will undergo pre-operative evaluation of their pain reporting accuracy ability in order to assess its relation to post-operative acute pain and analgesic consumption
  Interventions: Device: pain reporting accuracy

INTERVENTIONS:
Device: pain reporting accuracy — pain reporting accuracy will be assessed by the Focused Analgesia Selection Task (FAST) procedure. The FAST is based on recording a subject's pain reports in response to repeated administration of thermal noxious stimuli of various intensities, applied on the non-dominant arm with the Medoc® Thermal Sensory Analyzer II. The subjects will receive 1 of 7 designated temperatures (44°C, 45°C, 46°C, 47°C, 48°C, 49°C, and 50°C), each presented 7 times in a random block-ordered design (49 stimuli in total).

SUMMARY:
Pain is a subjective experience that differs in intensity from one person to another. Appropriate medical care relies on an accurate assessment of the patients' condition. However, when it comes to subjective assessment, accurate assessment is a challenge.

The most common tools used to estimate pain intensity depend on patient pain reports on a numerical pain scale (NPS) or a similar scales. Although these tools are widely used, there is a tendency to ignore the fact that the reliability and accuracy of pain reports are strongly influenced not only by the measuring instrument, but also by the person who uses it. A method has recently been developed to assess the accuracy of pain reports, and in a series of studies it has been found that the more accurate a person is in pain reports in response to stimulation,the smaller his placebo effect is .The aim of the study is to investigate whether assessing the accuracy of a person's pain reports can predict who will experience intensified post-operative pain and post-operative analgesic medications intake.The study will include 40 patients undergoing elective head & neck surgery. The study will be conducted prospectively and will include one pre-operative meeting to assess the accuracy of pain reports using the Focused Analgesia Selection Test (FAST). Patients will also complete pain-related psychological questionnaires during the session. In addition, post-operative pain measurements (NPS), and the use of pain relieving drugs (SOS) will be taken until release.

DETAILED DESCRIPTION:
Objectives and hypotheses: The purpose of this study is to examine whether pain reporting accuracy (as examined in the FAST test) predicts the intensity of acute post-operative pain and the consumption of pain-relieving drugs. The investigators hypothesize that the more accurate a person is in his pain reports, the more likely he will be to correlate postoperative pain and Analgesic drugs consumption.

The study population: The sample will include 40 subjects (men and women) who are about to undergo elective head & neck surgery in the Department of Otolaryngology.

Study design:

The institutional ethics committee of Carmel Medical Center approved the study protocol in accordance with the Helsinki Declaration, and written consent will be obtained from each subject before the beginning of the experiment. Participants will be enrolled into the study after meeting the inclusion criteria. The experiment will consist of one session, which will last about 45 minutes, during which the subject will undergo brief familiarization with the device, the stimulation and the scale in the study. Thereafter, all subjects will undergo the FAST procedure. Between the familiarization and the FAST, the subject will fill out pain-related personality questionnaires. From the moment of returning to the department after the surgery, the clinical follow-up will begin following pain reports and the consumption of pain-relieving drugs until the patient is released.

Psychophysical assessment: The contact-heat Q-sense system (Medoc, Ramat-Yishai, Israel) will be used to deliver the tonic heat stimulations applied by a 30 x 30 mm Peltier surface stimulator, which will be attached by Velcro straps to the volar surface of the forearm of the subject hand.

Familiarization: At the beginning of the experimental session, all subjects will undergo a short training in order to familiarize them with the device and with the sensations evoked by the painful stimulation, and to train them to report their perceived pain intensity using the numerical pain scale. The training will include exposure to three short contact-heat stimuli (44, 46.5, and 48°C), each lasting for 7 seconds from the time that the stimulation intensity reach the destination temperature. Subjects will be asked to report their pain on numerical pain scale (NPS) ranging from 0, denoting no pain, to 100, denoting the worst pain imaginable, induced by each stimulus.

Pain reporting accuracy assessment: Will be assessed by the FAST procedure. During the procedure, the thermode will be attached to the ventral surface of the subject's non-dominant arm and the temperature will be raised from a baseline of 32°C, peaks for 3 seconds at 1 of 7 designated temperatures (44°C, 45°C, 46°C, 47°C, 48°C, 49°C, and 50°C), and then decreased down to the baseline. Stimulus rate of rise and fall will be kept constant. Subjects will be asked to rate the peak pain intensity of each stimulus verbally using the NPS. Each temperature will be presented 7 times in a random block-ordered design (49 stimuli in total), with Inter-stimulus intervals of 20 seconds. The location of the thermode will be adjusted every 10 stimuli to minimize sensitization and/or habituation effects.

Evaluation of clinical variables: The clinical follow-up of patients begins from the moment the operation ends and continues until discharge (24-48 hours post-operation), and includes two measures:

1. Pain reports (NPS) - pain assessment at the time of analgesic medication consumption and an hour after administration of the drug, in addition to regular monitoring of every 6 hours during hospitalization. The reports will be documented by the nursing staff.
2. Follow-up after use of analgesic medications (according to the standard protocol + SOS medications including: Paracetamol IV, Optalgin PO, Oxycodone PO and Trimal IV).

Pain-related psychological questionnaires:

Pain sensitivity will be assessed by the Pain Sensitivity Questionnaire (PSQ). Dispositional optimism will be assessed by the Life Orientation Test-Revised (LOT-R).

Data analysis:

Data will be processed and analyzed using Excel , and SPSS® software version 23.

Descriptive statistics will be used to present demographic and baseline characteristics. Pain scores captured during the FAST procedure will be used to calculate 3 FAST outcomes as follows: 1) R2 will be calculated by using a power model regression. Disparity between the predicted function and actual scores could be a result of inaccuracy or unreliability. Close concordance between actual and predicted scores (higher R2) suggests greater accuracy and reliability. 2) Intraclass correlation coefficient (ICC) will be computed using a 2-way mixed model for the 7 presentations of each of the 7 intensity levels. An ICC score approaching 1.0 denotes a high degree of reliability or the agreement in responses to the same stimulus over several presentations. 3) The coefficient of variation (CoV) is the ratio of the standard deviation to the mean. The average CoV will be calculated as the mean of 7 CoVs, 1 at each stimulus level. Spearman's correlation between FAST outcome measures, NPS, analgesic consumption, PSQ and LOT-R will be calculated in order to assess relationships between pain reporting accuracy, clinical post-operative pain and pain-relates psychological measures. Exploring whether being identified as more painful patient in the acute post-operative phase (pro-nociceptive) could be predicted by pain reporting accuracy (as measures by FAST), and pain sensitivity (as assessed by PSQ) and optimism (as assessed by LOT-R) will be made by multivariate regression analyses.Statistical significance was defined as P≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Candidates to Head & Neck elective surgery

Exclusion Criteria:

* Presence of diagnosed psychiatric disorders, cognitive and /or neurological deficits;
* Use of analgesic, anti-depressants or anti-anxiolytics medications on a regular basis (except for oral contraceptives);
* Pregnancy.
* Inability to give informed consent, communicate, and understand the purpose and instructions of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in acute post-operative pain throughout the hospitalization period | From post-surgery recovery until discharge at specific time points: pain report (NPS) at the time of analgesic medication consumption, an hour after administration of the drug, in addition to regular monitoring of every 6 hours during hospitalization.
  Subjects will be asked to report their pain on numerical pain scale (NPS) ranging from 0, denoting "no pain", to 10, denoting "the worst pain imaginable".
Amount of analgesic drugs consumption I | From post-surgery recovery until discharge (24-48 hours after surgery)
  Quantification of the amount of analgesic drugs consumption will be performed by counting the number of times an SOS drug has been given. The SOS medications (beyond analgesic protocol) include Optalgin PO / Acamol IV / Oxycodone PO/ tramal IV.

SECONDARY OUTCOMES:
Amount of analgesic drugs consumption II | From post-surgery recovery until discharge (24-48 hours after surgery)
  Quantification of the amount of analgesic drugs consumption will be performed by conversion of opiates dosage into morphine units, out of the SOS medications that were taken.
Amount of analgesic drugs consumption III | From post-surgery recovery until discharge (24-48 hours after surgery)
  Quantification of the amount of analgesic drugs consumption will be performed by calculating the grams of NSAIDs consumption, out of the SOS medications that were taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel